CLINICAL TRIAL: NCT03831594
Title: Combining Physical Therapy With Vestibular Stimulation to Improve Postural Stability in Pusher's Syndrome
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: We were unable to recruit any suitable patients to this study
Sponsor: Imperial College London (Other)
Collaborators: Homerton University Hospital NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 222784
Record Dates: First submitted 2019-01-31; First posted 2019-02-06 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Pusher Syndrome
Keywords: stroke; galvanic vestibular stimulation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard Physiotherapy and Galvanic Vestibular Stimulation (Experimental): Standard physiotherapy concurrently with Galvanic Vestibular Stimulation for 45 minutes a day for two weeks (five days per week)
  Interventions: Device: Galvanic Vestibular Stimulation; Other: Standard Physiotherapy
- Standard Physiotherapy (Active Comparator): Standard Physiotherapy for 45 minutes a day for two weeks (five days per week)
  Interventions: Other: Standard Physiotherapy

INTERVENTIONS:
Device: Galvanic Vestibular Stimulation — Electrical current (under 1.5mA) applied to the mastoid processes to stimulate the balance organs in the inner ear
  Arms: Standard Physiotherapy and Galvanic Vestibular Stimulation
Other: Standard Physiotherapy — 45 minutes of standard physiotherapy treating impairments and functional problems
  Other Names: Standard Physical Therapy

SUMMARY:
The study is evaluating the effect of combining Galvanic Vestibular Stimulation (GVS) with standard Physiotherapy treatment in patients admitted to a neurological rehabilitation unit with Pusher syndrome (PS). Patients will be randomised to receive standard Physiotherapy treatment or standard treatment with GVS.

Perceived verticality data will also be collected and analysed on age-matched controls. This data will be used to compare these results with the patients with PS.

The investigators hypothesis that GVS and standard Physiotherapy treatment will lead to a greater improvement in functional ability and awareness of perceived verticality compared to standard Physiotherapy alone.

DETAILED DESCRIPTION:
Pusher syndrome (PS) can be described as disordered balance and orientation which causes patients to perceive they are in an upright position when in fact they are positioned towards their affected side. These patients use their unaffected limbs to 'push' themselves away from their unaffected side in an attempt to correct their perceived postural alignment. PS is a common disorder and can affect 16% of stroke patients.

Patients with PS have shown to take longer to improve in rehabilitation than non-PS patients and tend to stay in hospital for longer.

Galvanic Vestibular Stimulation (GVS) involves passing a small electrical current behind the ear to stimulate the vestibular system to in-turn cause the head and body to move.

ELIGIBILITY:
Pusher Inclusion Criteria:

* Identified hemiparetic neglect - identified PS from a stroke or acquired brain injury (using the Scale of Contraversive Pushing and The Burke Lateropulsion Scale)
* Consenting to participate in the trial

Pusher Exclusion Criteria:

* Severe cognitive impairment
* Receptive aphasia
* Medical co-morbidities
* Opthalamic impairment
* Vestibular impairment
* Peripheral neuropathy
* Also any contraindications to GVS including:

  * Brain metallic implants
  * Pacemakers
  * Recent brain surgery
  * Skull defect
  * Preceding epileptic seizures
  * Sensitive skin behind the ears.

Healthy volunteers inclusion criteria:

* 40 years old minimum age
* Consent to taking part in the trial

Healthy volunteers exclusion criteria:

* Vestibular impairment
* History of medical/psychiatric/neurological disorders
* Currently taking any psychoactive medication
* Drunk more than 3 units of alcohol in the past 24 hours

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2021-01-18 (Actual); Study Completion 2021-01-20 (Actual)

PRIMARY OUTCOMES:
Scale of Contraversive Pushing | Change from baseline, end of week 1 and end of week 2
  This is made up of 3 components: 1.The symmetry of spontaneous body posture (rated with 0, 0.25, 0.75, or 1 point. 1 = severe tilt, 0 = no tilt), 2. The use of non-paretic extremities (0, 0.5, or 1 point. 1 = performed spontaneously at rest), 3. The resistance to passive correction of the tilted posture (0 or 1 point. 1 = resistance occurs). For a diagnosis of Pusher Syndrome all 3 components need to be present.
The Burke Lateropulsion Scale | Change from baseline, end of week 1 and end of week 2
  Test of pushing. The score for each component is rated on a scale from 0 to 3 (0 to 4 for standing) and the score is based on the severity of resistance or the tilt angle when the patient begins to resist the passive movement. The score for diagnosis of Pusher behaviour is ≥2 points
Catherine Bergago Scale | Change from baseline, end of week 1 and end of week 2
  The Catherine Bergego Scale is a standardized checklist (10 everyday tasks) to detect presence and degree of neglect during observation of everyday life situations. The scale also provides a measure of neglect self-awareness (anosognosia).4 point rating scale indicating severity of neglect (0 = no neglect, 3 = severe neglect).
Mesulam's symbol cancellation test | Change from baseline, end of week 1 and end of week 2
  Mesulam's symbol cancellation test provides a measure of neglect, organisational process, and attention.
Berg Balance Scale | Change from baseline, end of week 1 and end of week 2
  14-item scale designed to measure balance of the older adult in a clinical setting. A five-point ordinal scale, ranging from 0-4. "0" indicates the lowest level of function and "4" the highest level of function. Score the LOWEST performance. Total Score = 56
Functional Impairment Measure | Change from baseline, end of week 1 and end of week 2
  18-item of physical, psychological and social function.The tool is used to assess a patient's level of disability as well as change in patient status in response to rehabilitation or medical intervention. Each item is scored on a 7 point ordinal scale, ranging from a score of 1 to a score of 7. The higher the score, the more independent the patient is in performing the task associated with that item.

SECONDARY OUTCOMES:
Subjective Visual Vertical | Change from baseline, end of week 1 and end of week 2
  Test of perceived visual vertical alignment
Subjective Postural Vertical | Change from baseline, end of week 1 and end of week 2
  Test of perceived postural vertical alignment
Subjective haptic vertical | Change from baseline, end of week 1 and end of week 2
  Test of perceived haptic vertical alignment

CONTACTS AND LOCATIONS:
Overall Officials: Diego Kaski, PhD, Principal Investigator — Imperial College London
Locations (1):
- Imperial College London, London, United Kingdom

REFERENCES:
- [Background] Baccini M, Paci M, Nannetti L, Biricolti C, Rinaldi LA. Scale for contraversive pushing: cutoff scores for diagnosing "pusher behavior" and construct validity. Phys Ther. 2008 Aug;88(8):947-55. doi: 10.2522/ptj.20070179. Epub 2008 Jul 10. PMID 18617579
- [Background] P. Azouvi (1996) Functional Consequences and Awareness of Unilateral Neglect: Study of an Evaluation Scale, Neuropsychological Rehabilitation, 6:2, 133-150, DOI: 10.1080/713755501
- [Background] Maggie J. Bailey, M. Jane Riddoch & Peter Crome (2004) Test-retest stability of three tests for unilateral visual neglect in patients with stroke: Star Cancellation, Line Bisection, and the Baking Tray Task, Neuropsychological Rehabilitation, 14:4, 403-419, DOI: 10.1080/09602010343000282
- [Background] Barra J, Marquer A, Joassin R, Reymond C, Metge L, Chauvineau V, Perennou D. Humans use internal models to construct and update a sense of verticality. Brain. 2010 Dec;133(Pt 12):3552-63. doi: 10.1093/brain/awq311. Epub 2010 Nov 19. PMID 21097492
- [Background] Day BL, Severac Cauquil A, Bartolomei L, Pastor MA, Lyon IN. Human body-segment tilts induced by galvanic stimulation: a vestibularly driven balance protection mechanism. J Physiol. 1997 May 1;500 ( Pt 3)(Pt 3):661-72. doi: 10.1113/jphysiol.1997.sp022051. PMID 9161984
- [Background] Fitzpatrick RC, Wardman DL, Taylor JL. Effects of galvanic vestibular stimulation during human walking. J Physiol. 1999 Jun 15;517 ( Pt 3)(Pt 3):931-9. doi: 10.1111/j.1469-7793.1999.0931s.x. PMID 10358131
- [Background] Karnath HO, Johannsen L, Broetz D, Ferber S, Dichgans J. Prognosis of contraversive pushing. J Neurol. 2002 Sep;249(9):1250-3. doi: 10.1007/s00415-002-0824-z. PMID 12242549
- [Background] Karnath HO, Broetz D. Understanding and treating "pusher syndrome". Phys Ther. 2003 Dec;83(12):1119-25. PMID 14640870
- [Background] Karnath HO. Pusher syndrome--a frequent but little-known disturbance of body orientation perception. J Neurol. 2007 Apr;254(4):415-24. doi: 10.1007/s00415-006-0341-6. Epub 2007 Mar 25. PMID 17385082
- [Background] Nakamura J, Kita Y, Yuda T, Ikuno K, Okada Y, Shomoto K. Effects of galvanic vestibular stimulation combined with physical therapy on pusher behavior in stroke patients: a case series. NeuroRehabilitation. 2014;35(1):31-7. doi: 10.3233/NRE-141094. PMID 24990006
- [Background] Parton A, Malhotra P, Husain M. Hemispatial neglect. J Neurol Neurosurg Psychiatry. 2004 Jan;75(1):13-21. PMID 14707298
- [Background] Perennou DA, Mazibrada G, Chauvineau V, Greenwood R, Rothwell J, Gresty MA, Bronstein AM. Lateropulsion, pushing and verticality perception in hemisphere stroke: a causal relationship? Brain. 2008 Sep;131(Pt 9):2401-13. doi: 10.1093/brain/awn170. Epub 2008 Aug 4. PMID 18678565
- [Background] Utz KS, Korluss K, Schmidt L, Rosenthal A, Oppenlander K, Keller I, Kerkhoff G. Minor adverse effects of galvanic vestibular stimulation in persons with stroke and healthy individuals. Brain Inj. 2011;25(11):1058-69. doi: 10.3109/02699052.2011.607789. Epub 2011 Aug 31. PMID 21879800